CLINICAL TRIAL: NCT02913625
Title: Retroclavicular Approach vs Infraclavicular Approach for Plexic Bloc Anesthesia of the Upper Limb: a Multi-centric Non-inferiority Randomised Controlled Trial
Brief Title: Retroclavicular Approach vs Infraclavicular Approach for Plexic Bloc Anesthesia of the Upper Limb
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Pablo Echave, Anesthesiologist, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MP-31-2017-1298
Record Dates: First submitted 2016-09-12; First posted 2016-09-26 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Hand Injury
Keywords: Brachial plexus; Regional anesthesia; Infraclavicular; Retroclavicular; Parasagittal; Upper limb surgery; Ultrasound guided block; Coracoid
MeSH Terms: conditions — Hand Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound guided retroclavicular block (Experimental): Patients assigned to this group will receive an ultrasound guided retroclavicular brachial plexus block
  Interventions: Other: Ultrasound guided retroclavicular block
- Ultrasound guided infraclavicular block (Active Comparator): Patients assigned to this group will receive an ultrasound guided infraclavicular brachial plexus block
  Interventions: Other: Ultrasound guided infraclavicular block

INTERVENTIONS:
Other: Ultrasound guided retroclavicular block — Ultrasound guided retroclavicular block for forearm or hand surgery
  Arms: Ultrasound guided retroclavicular block
Other: Ultrasound guided infraclavicular block — Ultrasound guided infraclavicular block for forearm or hand surgery
  Arms: Ultrasound guided infraclavicular block

SUMMARY:
Locoregional anesthesia provides several advantages over general anesthesia in terms of postoperative pain, decreased postoperative opioid needs and reduced recovery time for patients undergoing orthopaedic surgery.

For upper limb surgery, the coracoid infraclavicular brachial plexus block is generally preferred because of its simplicity and effectiveness but, needle visibility remains a challenge because of the angle between the ultrasound beam and the needle.

The retroclavicular approach for brachial plexus anesthesia requires an angle between the needle and the ultrasound beam that is less steep than the angle required to perform an infraclavicular coracoid block. This approach has already been proven effective and safe in the past.

The general objective is to provide a formal comparison between the retroclavicular approach and coracoid infraclavicular approach for brachial plexus anaesthesia. This study will delineate the differences between the two techniques.

DETAILED DESCRIPTION:
Investigators aim is to compare both techniques in terms of scanning time, needling time, total anesthesia time, needle visibility, block needle passes, block success and early and late complications. Investigators made the hypothesis that, while providing similar efficacy and better needle visualisation than coracoid infraclavicular block, performance time of retroclavicular block will not exceed the performance time of its comparator.

This study is designed as a prospective randomized non-inferiority trial. Two groups of non-consecutive patients will be randomly assigned to either retroclavicular or coracoid infraclavicular block. This study will be carried out in three different centres simultaneously.

The multicentre trial will be conducted in two university hospitals (Centre hospitalier universitaire de Sherbrooke [CHUS] Hôtel-Dieu/Fleurimont and Centre Hospitalier de l'Université Laval [CHUL] in Quebec city) and a community hospital (Cowansville). The third participating establishment, Brome-Missisquoi-Perkins hospital, is located in Cowansville, a peripheral city of 15,000 people.

ELIGIBILITY:
Inclusion Criteria:

* Elective or urgent surgery of the hand, wrist, forearm or elbow.
* Age >18 years old.
* ASA (American Society of Anesthesiologists) class 1, 2 and 3.
* Able to provide valid written consent.
* Minimum body weight of 50 kg, despite BMI

Exclusion Criteria:

* Patient refusal.
* Previous surgery or gross anatomical deformity of the clavicle.
* Systemic or local infection at needle entry point.
* Coagulopathy.
* Severe pulmonary condition.
* Local anaesthetic allergy.
* Pre-existing neurologic symptoms in the ipsilateral limb.
* Pregnancy.
* Surgical request of an indwelling catheter for post-operative analgesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2016-09; Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Time of block performance | Measured directly during the procedure with a chronometer. Time of performance is composed of imaging time and needling time
  The performance time corresponds to the sum of imaging time and needling time. It is expressed in minutes.
  Analysis of the primary outcome: performance time will be analyzed with a non-inferiority test of the averages, with the objective of finding that the experimental retroclavicular approach is no longer to perform than the coracoid infraclavicular approach.
  Subgroup analysis will be conducted to evaluate if higher body mass index influence (BMI) the outcomes, as the performance time, the needle visibility, the number of needle passes and the needle angle. Patient will be divided in two groups (higher and lower than the average BMI of all recruited patients) and analyzed according to their subgroup. If data is missing or if patient drop-out occurs, data will be analyzed with the intention-to-treat principle.

SECONDARY OUTCOMES:
Imaging time | Measured directly during the procedure with a chronometer.
  Corresponds to the time interval between contact of the US probe with the patient skin and the acquisition of a satisfactory image. It is expressed in minutes.
  The secondary outcomes will all be analyzed with superiority analysis. For continuous data or ordinal data with >8 categories, data will be compiled as average and standard deviation. If data is parametric, student T test will be used and if not, Mann-Whitney test will be used. For dichotomic data (block success, use of neurostimulation), Chi square or Fisher exact test will be used depending if all n>5 or if not, respectively. Finally, for ordinal data Chi square will be used if data is parametric and Mann-Whitney will be used otherwise
Needling time | Measured directly during the procedure with a chronometer.
  Corresponds to the time elapsed between the penetration of the skin with the needle until the complete removal of the needle from the tissues.
Time to sensory loss evaluated at 10, 20 and 30 minutes after procedure | Blind assistant evaluates the loss of sensibility in 5 precise nerve territories, 10, 20 and 30 minutes after the block.
  Sensory loss will be assessed in the territory of the radial (lateral aspect of the dorsum of the hand), median (volar aspect of the index), ulnar (volar aspect of the fifth finger), musculocutaneous (lateral aspect of the forearm), and medial cutaneous nerve of the forearm (medial aspect of the forearm) distributions using a 3-point score, where 0 = normal sensation, 1 = diminished sensation to pinpricks (hypoesthesia), and 2 = loss of sensation to pinpricks (analgesia). The sum of five scores on a maximum of 10 will be the sensory loss final score. An independent, blinded, research assistant will complete the sensory assessment at 10, 20 and 30 minutes after procedure
Time to motor blockade evaluated at 10, 20 and 30 minutes after procedure | Blind assistant evaluates the loss of motor function in four muscular groups at 10, 20 and 30 minutes after the block.
  Motor function will be tested (0 = normal strength, 1 = weakness, 2 = paralysis) for the radial (wrist extension), median (thumb-fifth finger opposition), ulnar (fifth finger abduction), and musculocutaneous (elbow flexion) nerves. The sum of the four scores on a maximum of 8 will be the motor block final score. An independent, blinded, research assistant will complete the motor assessment at 10, 20 and 30 minutes after procedure
Success of plexus block | Success is defined at end of surgery for which block was done, generally within 1 to 3 hours after block is performed
  Success is defined as the completion of surgery without the need for additional local anesthetics infiltration, intravenous narcotics, or general anesthesia. However, light sedation is allowed if deemed necessary by the anesthesiologist. Light sedation includes midazolam 1 to 4 mg intravenously, fentanyl up to 1 mcg/kg. A minimum sensory score of 9/10 will be necessary to proceed to surgery without additional local anesthetics infiltration. Patients with an overall sensory score less than 9/10 at 30 minutes will be offered general anesthesia or supplemental blocks.
Total anesthesia time | Intraoperative
  Measured in minutes and defined as the sum of performance time and time to achieve a minimum sensory score of 9/10. It is the time for readiness for surgery.
Number of needle passes | Number of needle passes required during procedure.
  Defined as a unit of 1,2,3, etc. The number of times the block needle will have to be realigned at the skin in order to achieve its final positioning goal under the axillary artery.
Needle visualization | Assessed one week after study completion
  Procedures will be videotaped and reviewed simultaneously after study completion by 2 independent anesthesiologists skilled in US-guided regional anesthesia using a 5-point Likert scale to rate needle visibility (1=very poor,2=poor,3=fair,4=good,5=very good). Needle visibility will be evaluated twice. First, for the retroclavicular approach, assessment will be done when needle tip is seen 1cm after crossing the clavicle acoustic shadowing. For the coracoid infraclavicular approach, the first assessment will be at a needle tip depth of 1 cm. Second needle visibility assessment will be immediately before local anesthetic injection when block needle is positioned under axillary artery (when the visibility is theoretically optimized)
Needle angle | Assessed one week after study completion
  Using the same videotape that investigators used for the evaluation of the needle visibility, the angle between the needle and the upper side of the ultrasound image will be noted. It will be a continuous outcome ranging from 0 to 90 degrees.
Neurostimulation use | Assessed during the block
  Neurostimulation is accepted if needed. However, its use other than for safety sentinel (defined by <0,3 mA) will be recorded for subsequent analysis. It will be a dichotomic outcome.
Pain during the procedure | Patients will be asked to report the level of discomfort they felt during the procedure
  Immediately after block completion, patients will be asked to rate their discomfort associated with the procedure using a 10-cm visual analogue scale (0 = no pain, 10 = worst pain imaginable) by an independent and blinded outcome assessor.
Early and late complications: | Assessed during each block and again at 48 hours after the block
  The incidence of needle-induced paresthesia, vascular puncture, Horner syndrome, dyspnea, and symptoms of local anesthetics toxicity will be noted. All patients will be contacted 48 hours after surgery to ask for any delayed complications, such as dyspnea, paresthesia, weaknesses, pain at the puncture site, hematoma.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Echave, M.D., Principal Investigator — Université de Sherbrooke
Locations (2):
- Canada (2):
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
  - Centre Hospitalier de l'Université Laval [CHUL], Québec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hadzic A, Arliss J, Kerimoglu B, Karaca PE, Yufa M, Claudio RE, Vloka JD, Rosenquist R, Santos AC, Thys DM. A comparison of infraclavicular nerve block versus general anesthesia for hand and wrist day-case surgeries. Anesthesiology. 2004 Jul;101(1):127-32. doi: 10.1097/00000542-200407000-00020. PMID 15220781
- [Background] Bruce BG, Green A, Blaine TA, Wesner LV. Brachial plexus blocks for upper extremity orthopaedic surgery. J Am Acad Orthop Surg. 2012 Jan;20(1):38-47. doi: 10.5435/JAAOS-20-01-038. PMID 22207517
- [Background] Chin KJ, Alakkad H, Adhikary SD, Singh M. Infraclavicular brachial plexus block for regional anaesthesia of the lower arm. Cochrane Database Syst Rev. 2013 Aug 28;2013(8):CD005487. doi: 10.1002/14651858.CD005487.pub3. PMID 23986434
- [Background] Lopez-Morales S, Moreno-Martin A, Leal del Ojo JD, Rodriguez-Huertas F. [Ultrasound-guided axillary block versus ultrasound-guided infraclavicular block for upper extremity surgery]. Rev Esp Anestesiol Reanim. 2013 Jun-Jul;60(6):313-9. doi: 10.1016/j.redar.2013.02.012. Epub 2013 May 15. Spanish. PMID 23684374
- [Background] Vermeylen K, Engelen S, Sermeus L, Soetens F, Van de Velde M. Supraclavicular brachial plexus blocks: review and current practice. Acta Anaesthesiol Belg. 2012;63(1):15-21. PMID 22783706
- [Background] Trehan V, Srivastava U, Kumar A, Saxena S, Singh CS, Darolia A. Comparison of two approaches of infraclavicular brachial plexus block for orthopaedic surgery below mid-humerus. Indian J Anaesth. 2010 May;54(3):210-4. doi: 10.4103/0019-5049.65362. PMID 20885866
- [Background] Minville V, Asehnoune K, Chassery C, N'Guyen L, Gris C, Fourcade O, Samii K, Benhamou D. Resident versus staff anesthesiologist performance: coracoid approach to infraclavicular brachial plexus blocks using a double-stimulation technique. Reg Anesth Pain Med. 2005 May-Jun;30(3):233-7. doi: 10.1016/j.rapm.2005.01.009. PMID 15898025
- [Background] de Gusmao LC, Lima JS, Ramalho Jda R, Leite AL, da Silva AM. Evaluation of brachial plexus fascicles involvement on infraclavicular block: unfixed cadaver study. Braz J Anesthesiol. 2015 May-Jun;65(3):213-6. doi: 10.1016/j.bjane.2014.06.010. Epub 2015 Feb 17. PMID 25925034
- [Background] Tsui, B.C.-H., Atlas of ultrasound and nerve stimulation-guided regional anesthesia. 2007: New York : Springer.
- [Background] Hebbard P, Royse C. Ultrasound guided posterior approach to the infraclavicular brachial plexus. Anaesthesia. 2007 May;62(5):539. doi: 10.1111/j.1365-2044.2007.05066.x. No abstract available. PMID 17448088
- [Background] Charbonneau J, Frechette Y, Sansoucy Y, Echave P. The Ultrasound-Guided Retroclavicular Block: A Prospective Feasibility Study. Reg Anesth Pain Med. 2015 Sep-Oct;40(5):605-9. doi: 10.1097/AAP.0000000000000284. PMID 26222346
- [Background] Beh ZY, Hasan MS, Lai HY, Kassim NM, Md Zin SR, Chin KF. Posterior parasagittal in-plane ultrasound-guided infraclavicular brachial plexus block-a case series. BMC Anesthesiol. 2015 Jul 21;15:105. doi: 10.1186/s12871-015-0090-0. PMID 26194896
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Background] Tran DQ, Clemente A, Tran DQ, Finlayson RJ. A comparison between ultrasound-guided infraclavicular block using the "double bubble" sign and neurostimulation-guided axillary block. Anesth Analg. 2008 Sep;107(3):1075-8. doi: 10.1213/ane.0b013e31817ef259. PMID 18713932
- [Background] Yazer MS, Finlayson RJ, Tran DQ. A randomized comparison between infraclavicular block and targeted intracluster injection supraclavicular block. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):11-5. doi: 10.1097/AAP.0000000000000193. PMID 25478758
- [Derived] Blanco AFG, Laferriere-Langlois P, Jessop D, D'Aragon F, Sansoucy Y, Albert N, Tetreault P, Echave P. Retroclavicular vs Infraclavicular block for brachial plexus anesthesia: a multi-centric randomized trial. BMC Anesthesiol. 2019 Oct 27;19(1):193. doi: 10.1186/s12871-019-0868-6. PMID 31656165
- [Derived] Langlois PL, Gil-Blanco AF, Jessop D, Sansoucy Y, D'Aragon F, Albert N, Echave P. Retroclavicular approach vs infraclavicular approach for plexic bloc anesthesia of the upper limb: study protocol randomized controlled trial. Trials. 2017 Jul 21;18(1):346. doi: 10.1186/s13063-017-2086-1. PMID 28732521